CLINICAL TRIAL: NCT01470885
Title: the Influence of Glucose to the Prognosis of Patients of Acute Pancreatitis
Brief Title: Relation of Glucose and Acute Pancreatitis
Acronym: ROGAAP
Status: Completed | Type: Observational
Sponsor: Huashan Hospital (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, xiaolong zhao, endocrinology department, Huashan Hospital
Other Study IDs: zsdxxhnk20110707
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Acute Pancreatitis
Keywords: glucose; prognosis; glycated hemoglobin
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- glucose value: glucose value

SUMMARY:
Acute pancreatitis (AP) is an acute inflammatory disease of the pancreas which can lead to a systemic inflammatory response syndrome with significant morbidity and mortality in 20% of patients. Part of endocrine function of pancreas would be affected in AP. Stress hyperglycemia would explode at acute phase. So the investigators decide to follow up and observe 200 cases of patients with acute pancreatitis, determining of blood sugar, blood amylase, hemoglobin and glycosylated hemoglobin level. At last, using ROC curve method to identify the die cutting between blood glucose level and acute pancreatitis, and makes analysis of the diagnostic value.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) is an acute inflammatory disease of the pancreas which can lead to a systemic inflammatory response syndrome with significant morbidity and mortality in 20% of patients. Part of endocrine function of pancreas would be affected in AP. Stress hyperglycemia would explode at acute phase. There are two reasons. One is because that sympathetic hyperactivity makes glucagon elevated. Secondary, microcirculation disorder makes pancreas edema, ischemia and necrosis, affecting secretion and excretion of insulin. In severe acute pancreatitis, there may be ketoacidosis. Many scoring systems for predicting prognosis of severe acute pancreatitis also contains glucose values, such as the Ranson scoring system and the Glascow scoring system. On the other hand, Type 2 diabetes has become a global pandemic disease. Most of patients of type 2 diabetes are obese, who easily complicated gallstone disease and hypertriglyceridemia. All of above could be the risk factors for acute pancreatitis. Our initial small sample research also suggests undiagnosed diabetes patients whose glucose value elevated is significantly worse than the known diabetic patients. Therefore, the investigators believe that glucose directly affects the prognosis of AP. So the investigators decide to follow up and observe 1000 cases of patients with acute pancreatitis, determining of blood sugar, blood amylase, hemoglobin and glycosylated hemoglobin level. At last, using ROC curve method to identify the die cutting between blood glucose level and acute pancreatitis, and makes analysis of the diagnostic value.

ELIGIBILITY:
Inclusion Criteria:

patients that newly diagnosed as acute pancreatitis.

Exclusion Criteria:

exclude other acute abdomen, such as peptic ulcer with perforation, mesenteric arterial embolism or ruptured ectopic pregnancy.

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2011-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
motability | motability
  motability after acute pancreatitis

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaolong Zhao, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Zhao X, Chang Mei H, Chen L, Jiang L, He M, Chen J, Hu Z, Ye H, Hu H, Zhou L, Li Y, Hu R. An increased level of haemoglobin A1C predicts a poorer clinical outcome in patients with acute pancreatitis. Clin Endocrinol (Oxf). 2012 Aug;77(2):241-5. doi: 10.1111/j.1365-2265.2011.04252.x. PMID 21988175